CLINICAL TRIAL: NCT04076020
Title: Mobile Health Intervention for Rural Atrial Fibrillation
Brief Title: Atrial Fibrillation Health Literacy and Information Technology Trial in Rural Pennsylvania Counties
Acronym: AFibLITT_R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Northeastern University (Other); Boston University (Other)
Responsible Party: Principal Investigator, Jared W Magnani, MD, MSc, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY19050386; R01HL143010 (NIH)
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Familial Atrial Fibrillation; Arrhythmia, Cardiac; Heart Diseases; Pathologic Processes
Keywords: Adherence; Health Literacy; quality of life
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Pathologic Processes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive the relational agent and the AliveCor Kardia for use for 120 days. Participants are directed to use these interventions daily.
  Interventions: Behavioral: Relational agent/AliveCor Kardia - Intervention
- Usual Care (Active Comparator): Receive a brochure on atrial fibrillation that is published by the American Heart Association and a smartphone with the WebMD application.
  Participants are directed to use the WebMD application as often as they would like.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Relational agent/AliveCor Kardia - Intervention — Use of the relational agent and Kardia daily for 120 days.
  Arms: Intervention
Behavioral: Usual Care — Use of the WebMD app daily for 120 days.
  Arms: Usual Care

SUMMARY:
Atrial fibrillation (AF) is a highly prevalent, morbid condition. Anticoagulation to prevent thromboembolic strokes is a foremost priority in AF but adherence is challenging for patients and lapses in anticoagulation are common. Chronic disease self-management (CDSM) is a recognized program to enhance self-efficacy and improve adherence, quality of life, and patient-centered health outcomes. Rural patients with AF experience increased vulnerability to adverse outcomes due to geographic and social isolation, poor health care access, and limited health literacy. This study uses an innovative, scalable CDSM intervention to improve anticoagulation adherence in rural patients with AF.

DETAILED DESCRIPTION:
This is a randomized clinical trial to evaluate the effect of an embodied conversational agent (ECA) on health outcomes in people with atrial fibrillation. The study will enroll 264 patients who reside in rural, Western Pennsylvania who have atrial fibrillation. Participants will be randomized to the intervention or usual care. Intervention participants will receive a contemporary mobile phone, commonly known and referred to herein as a smartphone, with a relational agent, which simulates conversation and provides coaching, guidance, and assistance with chronic disease self-management. In addition participants will receive an FDA-approved instrument for heart rate and rhythm monitoring, which is named the "AliveCor KardiaMobile" device (herein referred to as the AliveCor Kardia), that pairs with the relational agent. Usual care participants will receive a smartphone as well, which will have the general health application called "WebMD." The intervention will last 4 months and participants will have visits at baseline, 4, 8 and 12 months. The study will evaluate the improvement in adherence to anticoagulation, quality of life, and health care utilization resulting from the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, age ≥21;
2. Diagnosis of AF, identified from the electronic health record (EHR) problem list and confirmed by 2 or more reports of AF from separate monitoring events at least 2 weeks apart (CG, Holter or event monitor);
3. Prescribed use of warfarin or direct-acting oral anticoagulant (DOAC) for AF stroke prevention;
4. English-speaking well enough to participate in informed consent and this study;
5. No plans to relocate from the area within 12 months of enrollment.

Exclusion Criteria:

1. Conditions other than AF that require anticoagulation, such as mechanical prosthetic valve, deep vein thrombosis, or pulmonary embolism;
2. History of pulmonary vein isolation or foreseen pulmonary vein isolation;
3. History of atrioventricular (AV) nodal ablation or foreseen AV nodal ablation;
4. Heart failure necessitating hospital admission ≤3 months prior to study inclusion;
5. Acute coronary syndrome (defined as at least 2 of the following: chest pain, ischemic electrocardiographic changes, or troponin ≥0.1 ng/mL) ≤3 months prior to study inclusion;
6. Untreated hyperthyroidism or ≤3 months euthyroidism before inclusion;
7. Foreseen pacemaker, internal cardioverter defibrillator, or cardiac resynchronization therapy;
8. Cardiac surgery ≤3 months before inclusion;
9. Planned cardiac surgery;
10. Presence of non-cardiovascular conditions likely to be fatal within 12 months (e.g., cancer);
11. Inability to comprehend the study protocol, defined as failing to answer correctly a set of questions on orientation and short-term memory during the consent process.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared W. Magnani, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will share individual participant data that underlie the results reported in the study's central manuscripts after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Such data will be available beginning 9 months and ending 36 months following publication of the main manuscripts resulting from this clinical trial.
Access Criteria: Data will be made available to those investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Proposals may be submitted up to 36 months following article publication. Applicants requesting access to the data will be responsible for the minimal administrative costs to provide the data set.

REFERENCES:
- [Derived] Mann HK, Streiff M, Schultz KC, Halpern DV, Ferry D, Johnson AE, Magnani JW. Rurality and Atrial Fibrillation: Patient Perceptions of Barriers and Facilitators to Care. J Am Heart Assoc. 2023 Nov 7;12(21):e031152. doi: 10.1161/JAHA.123.031152. Epub 2023 Oct 27. PMID 37889198
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at numerous University of Pittsburgh Medical Center (UPMC) sites located in rural Pennsylvania counties. The first participant was enrolled on January 8th, 2020 and the last participant was enrolled in March 2022.
Groups:
- Intervention: ECA/Kardia: Participants received the relational agent and the AliveCor Kardia to use for 120 days.
  Participants were directed to use the relational agent and AliveCor Kardia daily.
  Relational agent/AliveCor Kardia - Intervention Group: Use of the relational agent and Kardia daily for 120 days.
- Control: WebMD: Participants received a brochure on atrial fibrillation that is published by the American Heart Association and a smartphone with the WebMD application.
  Participants were directed to use the WebMD application as often as they would like.
  Usual Care: Use of the WebMD app daily for 120 days.
Period: Overall Study
Arm/Group | Intervention: ECA/Kardia | Control: WebMD
Started | 135 | 135
Completed | 119 | 121
Not Completed | 16 | 14
Not completed — Death | 4 | 6
Not completed — Withdrawal by Subject | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm: Participants received the relational agent and the AliveCor Kardia to use for 120 days.
  Participants were directed to use the relational agent and AliveCor Kardia daily.
  Relational agent/AliveCor Kardia - Intervention Group: Use of the relational agent and Kardia daily for 120 days.
- Usual Care Arm: Participants received a brochure on atrial fibrillation that is published by the American Heart Association and a smartphone with the WebMD application.
  Participants were directed to use the WebMD application as often as they would like.
  Usual Care: Use of the WebMD app daily for 120 days.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Usual Care Arm | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73.6 [66.8 to 78.8] | 72.7 [67.9 to 78.5] | 73.1 [67.5 to 78.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 83 | 163
  Male | 55 | 52 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 131 | 130 | 261
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 129 | 128 | 257
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Anticoagulant medication used for stroke prevention [Count of Participants; unit: Participants] — Participant receipt of oral medication for thromboembolic stroke prevention, classified as either warfarin or direct acting oral anticoagulant.
  Participants
    Warfarin | 22 | 22 | 44
    Direct acting oral anticoagulant | 113 | 113 | 226
Education [Count of Participants; unit: Participants]
  High school, vocational or trade school or less | 70 | 58 | 128
  Some College or associate degree | 39 | 37 | 76
  College (Bachelors or higher) | 26 | 40 | 66
Employment Status [Count of Participants; unit: Participants]
  Currently Working, Part-time or Full-time | 20 | 15 | 35
  Not Currently Working | 11 | 13 | 24
  Retired | 104 | 107 | 211
Marital Status [Count of Participants; unit: Participants]
  Single, not married | 7 | 5 | 12
  Married or living as married | 86 | 95 | 181
  Separated or divorced | 18 | 10 | 28
  Widowed | 24 | 25 | 49
Cohabitation [Count of Participants; unit: Participants]
  Resides with others | 86 | 95 | 181
  Resides alone | 49 | 40 | 89
Housing [Count of Participants; unit: Participants]
  Renting | 17 | 14 | 31
  Buying, and Paying mortgage | 22 | 25 | 47
  Own | 92 | 93 | 185
  Neither own nor pay rent | 4 | 2 | 6
  Prefer not to respond | 0 | 1 | 1
Housing ownership status [Count of Participants; unit: Participants]
  Ownership | 92 | 93 | 185
  Rent or other status | 43 | 42 | 85
Hypertension [Count of Participants; unit: Participants]
  Yes | 117 | 117 | 234
  No | 18 | 18 | 36
Smoking [Count of Participants; unit: Participants]
  Never Smoke | 62 | 74 | 136
  Current Smoker | 12 | 5 | 17
  Past Smoker | 61 | 56 | 117
Alcohol consumption, heavy [Count of Participants; unit: Participants] — Dichotomous indication of "Heavy weekly drinking," determined by self-report. Heavy alcohol consumption determined in women, 8 or more drinks/week and in men, 15 or more drinks/week
  Participants
    Yes | 5 | 5 | 10
    No | 130 | 130 | 260
History of any cardioversion [Count of Participants; unit: Participants] — History of treatment with electrical cardioversion and/or pharmacologic cardioversion. Some participants reported undergoing both electrical and pharmacologic cardioversion.
  Participants
    Yes | 43 | 37 | 80
    No | 92 | 98 | 190
Electrical Cardioversion [Count of Participants; unit: Participants] — History of cardioversion performed by administration of electrical therapy.
  Participants
    Yes | 40 | 35 | 75
    No | 95 | 100 | 195
Pharmacologic cardioversion [Count of Participants; unit: Participants] — History of cardioversion performed by administration of pharmacologic therapy
  Participants
    Yes | 5 | 2 | 7
    No | 130 | 133 | 263
Health Literacy [Count of Participants; unit: Participants] — The Newest Vital Sign tool was used to assess health literacy. Scores range from 0 to 6, with limited limited health literacy defined by a score of 0 to 3 and adequate health literacy by a sore of 4 to 6.
  Participants
    Limited Health Literacy | 63 | 62 | 125
    Adequate Health Literacy | 72 | 73 | 145
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index recorded directly from the electronic health record.
  kg/m^2 | 32.8 (8.1) | 33.5 (8.7) | 33.1 (8.4)
AF History [Mean (Standard Deviation); unit: years] — Duration in years
  years | 5.8 (6.7) | 7.0 (8.7) | 6.4 (7.7)
AF Effect on Quality-of-Life questionnaire (AFEQT) [Mean (Standard Deviation); unit: units on a scale] — AF Effect on Quality-of-Life questionnaire (AFEQT)
  Overall score and individual domain scores at baseline.
  Scoring: Scores for the overall score and each subscale range from 0-100. A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered).
  units on a scale
    Overall | 75.1 (15.1) | 73.7 (17.0) | 74.4 (16.1)
    Symptoms | 85.5 (15.0) | 83.5 (17.1) | 84.5 (16.1)
    Daily activities | 66.0 (23.6) | 67.1 (25.0) | 66.6 (24.2)
    Treatment concern | 80.4 (16.6) | 76.1 (19.1) | 78.2 (18.0)
    Treatment Satisfaction: How well treatment controls symptoms | 82.6 (17.5) | 79.0 (18.9) | 80.8 (18.3)
    Treatment satisfaction: Relief of symptoms | 81.0 (19.0) | 77.7 (21.6) | 79.3 (20.4)
Patient-Reported Outcomes Measurement Information System (PROMIS-29) [Median (Inter-Quartile Range); unit: units on a scale] — The Patient-Reported Outcomes Measurement Information System (PROMIS-29) assesses 7 domains with 4 questions each with scores transformed using a T-score such that scores have a mean of 50 and standard deviation of 10 in a referent population. Domains are: physical function; depression and sadness; pain interference; satisfaction with participation in social roles and activities; fatigue; anxiety and fear; and sleep disturbance. Higher scores indicate worse or more severe depression, pain, fatigue, anxiety/sleep domains, while better health for the physical function and satisfaction domains.
  units on a scale
    Physical function | 41.7 [36.0 to 47.6] | 42.9 [36.6 to 48.2] | 41.8 [36.4 to 48.2]
    Depression and sadness | 41.0 [41.0 to 52.1] | 48.9 [41.0 to 55.4] | 48.9 [41.0 to 54.1]
    Pain interference | 53.9 [41.6 to 60.0] | 55.7 [41.6 to 61.3] | 54.8 [41.6 to 61.3]
    Satisfaction with participation in social roles and activities | 53.9 [41.6 to 60.0] | 55.7 [41.6 to 61.3] | 54.8 [41.6 to 61.3]
    Fatigue | 51.0 [46.0 to 55.2] | 51.9 [48.6 to 60.7] | 51.0 [46.0 to 58.7]
    Anxiety and fear | 48.2 [40.3 to 55.2] | 51.4 [40.3 to 57.5] | 50.4 [40.3 to 56.0]
    Sleep disturbance | 51.0 [44.3 to 55.8] | 50.8 [44.2 to 55.8] | 51.0 [44.2 to 55.8]
Self-reported adherence [Count of Participants; unit: Participants] — Self-reported daily adherence to oral anticoagulation dichotomized as adherent or non-adherent. Three-item instrument each scaled 1-5. Individuals reporting 1 for all items classified as adherent; any individual reporting 2 or higher on any item classified as non-adherent.
  Participants
    Adherent | 120 | 119 | 239
    Non-adherent | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days Covered
Description: Proportion of Days Covered (PDC), obtained from collection of electronic prescription and pharmacy fill data, and defined as the proportion of availability of medication for the period of interest. PDC range is 0 to 1.00 with higher values indicating greater proportion of days with medication as indicated by pharmacy records.
Time Frame: 12 months
Population: Initial data set included 270 participants. 7 cases of no pharmacy data, 12 cases with start date after end date, and 1 case where one fill was available before randomization. PDC was calculated for 250 participants.
Measure: Median (Inter-Quartile Range); unit: Proportion of days covered
Groups:
- Intervention: Participants received the relational agent and the AliveCor Kardia to use for 120 days.
  Participants were directed to use the relational agent and AliveCor Kardia daily.
- Usual Care: Participants received a brochure on atrial fibrillation that is published by the American Heart Association and a smartphone with the WebMD application.
  Participants were directed to use the WebMD application as often as they would like.
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 124 | 126
Proportion of days covered | .97 [0.89 to 1.00] | 0.97 [0.92 to 1.00]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Proportion of days covered (PDC) at 12 months. A sample size of 119 in each study arm enabled us to detect a minimum difference in PDC of 11.7% with 85% power (assuming a standard deviation=30%). Our power calculations assume use of 2-sided tests with 0.05 significance level; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney) — Results presented from Wilcoxon-Mann-Whitney test with PDC as the dependent variable
Statistical Analysis 2: Comparison: Intervention vs Usual Care; Proportion of days covered (PDC) analyzed as a binary variable with optimal adherence determined as ≥0.80) variables using logistic regression and adjustment for trial stratification factors. Our power calculations assume use of 2-sided tests with 0.05 significance level; Test type: Superiority; p < 0.05, Regression, Logistic

2. Primary Outcome: Self-reported Adherence
Description: Self-reported adherence to oral anticoagulation. 3-item instrument with range 1-5 such that lower scores indicate more frequent medication adherence. Here the score is dichotomized by classifying participants reporting 1 for all three items as adherent and those that reported ≥ 2 on any item as non-adherent.
Time Frame: 4, 8, and 12 months
Population: Intervention 4-month: n=117 (11 withdrawals [w/d], 1 death; 4 discontinued [d/c] oral anticoagulation [OAC]; 2 missed visit) 8-month: n=114 (total 12 w/d, 4 deaths; 3 d/c OAC; 2 missed visit) 12-month: n=114 (total 12 w/d, 4 deaths, 5 d/c OAC)
  Control 4-month: n=121 (8 w/d, 4 deaths; 1 d/c OAC; 1 missed visit) 8-month: n=118 (total 8 w/d, 6 deaths; 3 d/c OAC) 12-month: n=115 (total 8 w/d, 6 deaths; 4 d/c OAC; 2 missed visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 135 | 135
Participants
  Adherence-4 Months: number analyzed (Participants) | 117 | 121
  Adherence-4 Months: Adherent | 112 | 107
  Adherence-4 Months: Non-adherent | 5 | 14
  Adherence-8 Months: number analyzed (Participants) | 114 | 118
  Adherence-8 Months: Adherent | 106 | 93
  Adherence-8 Months: Non-adherent | 8 | 25
  Adherence-12 Months: number analyzed (Participants) | 114 | 115
  Adherence-12 Months: Adherent | 104 | 98
  Adherence-12 Months: Non-adherent | 10 | 17
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Difference in self-reported adherence reported across baseline, 4-, 8-, and 12-month visits using generalized estimating equations and adjusted for trial stratification factors; Test type: Superiority; p < 0.05, Regression, Logistic

3. Secondary Outcome: Atrial Fibrillation Effect on Quality of Life (AFEQT)
Description: The AFEQT is a widely used measure of atrial fibrillation-specific health-related quality of life which consists of a global score and 4 domains (symptoms, daily activities, treatment concerns, and treatment satisfaction). Overall or subscale scores range from 0-100 with higher scores indicating superior health-related quality of life in AF. A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered).
Time Frame: 4, 8, and 12 months
Population: Intervention arm:
  4-month visit, n=121 (11 withdrawals, 1 death; 2 missed this visit) 8-month visit, n=117 (total 12 withdrawals, 4 deaths; 2 missed this visit) 12-month visit, n=119 (no additional withdrawals, no additional deaths, no missed visit)
  Control arm:
  4-month visit, n=122 (8 withdrawals, 4 deaths; 1 missed this visit) 8-month visit, n=121 (total 6 deaths; no missed this visit) 12-month visit, n=119 (no additional withdrawals, no additional deaths; 2 missed this visit)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 135 | 135
score on a scale
  Overall Score : 4-month: number analyzed (Participants) | 121 | 122
  Overall Score : 4-month | 77.8 [60.2 to 88.0] | 75.9 [63.0 to 90.7]
  Overall Score : 8-month: number analyzed (Participants) | 117 | 121
  Overall Score : 8-month | 81.5 [63.9 to 92.6] | 79.6 [66.7 to 93.5]
  Overall Score: 12-month: number analyzed (Participants) | 119 | 119
  Overall Score: 12-month | 80.6 [63.9 to 88.9] | 77.8 [62.0 to 90.7]
  Symptoms : 4-month: number analyzed (Participants) | 121 | 122
  Symptoms : 4-month | 87.5 [70.8 to 95.8] | 91.7 [75.0 to 100.0]
  Symptoms : 8-month: number analyzed (Participants) | 117 | 121
  Symptoms : 8-month | 91.7 [75.0 to 100.0] | 91.7 [79.2 to 100.0]
  Symptoms : 12-month: number analyzed (Participants) | 119 | 119
  Symptoms : 12-month | 91.7 [70.8 to 100.0] | 91.7 [75.0 to 100.0]
  Daily Activities : 4-month: number analyzed (Participants) | 121 | 122
  Daily Activities : 4-month | 70.8 [41.7 to 85.4] | 68.8 [50.0 to 89.6]
  Daily Activities : 8-month: number analyzed (Participants) | 117 | 121
  Daily Activities : 8-month | 75.0 [54.2 to 91.7] | 75.00 [54.2 to 93.8]
  Daily Activities : 12-month: number analyzed (Participants) | 119 | 119
  Daily Activities : 12-month | 70.8 [47.9 to 87.5] | 72.9 [45.8 to 89.6]
  Treatment Concern : 4-month: number analyzed (Participants) | 121 | 122
  Treatment Concern : 4-month | 83.3 [69.4 to 97.2] | 83.3 [66.7 to 97.2]
  Treatment Concern : 8-month: number analyzed (Participants) | 117 | 121
  Treatment Concern : 8-month | 88.9 [72.2 to 97.2] | 86.1 [69.4 to 94.2]
  Treatment Concern : 12-month: number analyzed (Participants) | 119 | 119
  Treatment Concern : 12-month | 88.9 [69.4 to 97.2] | 86.1 [69.4 to 94.4]
  Satisfaction: Relief of Symptoms: 4-month: number analyzed (Participants) | 121 | 122
  Satisfaction: Relief of Symptoms: 4-month | 83.0 [66.7 to 100.0] | 83.0 [66.7 to 100.0]
  Satisfaction: Relief of Symptoms: 8-month: number analyzed (Participants) | 117 | 121
  Satisfaction: Relief of Symptoms: 8-month | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0]
  Satisfaction: Relief of Symptoms: 12-month: number analyzed (Participants) | 119 | 119
  Satisfaction: Relief of Symptoms: 12-month | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0]
  Satisfaction: Control of Symptoms: 4-month: number analyzed (Participants) | 121 | 122
  Satisfaction: Control of Symptoms: 4-month | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0]
  Satisfaction: Control of Symptoms: 8-month: number analyzed (Participants) | 117 | 121
  Satisfaction: Control of Symptoms: 8-month | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0]
  Satisfaction: Control of Symptoms: 12-month: number analyzed (Participants) | 119 | 119
  Satisfaction: Control of Symptoms: 12-month | 83.3 [66.7 to 100.0] | 83.3 [66.7 to 100.0]

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)-29
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 assesses 7 domains (physical function; depression and sadness; pain interference; satisfaction with participation in social roles and activities; fatigue; anxiety and fear; sleep disturbance), 4 questions each, and Pain Intensity with a single item. The 7 domain scores are transformed using a T-score with a mean of 50, standard deviation of 10, in a referent population. Higher scores indicate worse health for the depression, pain, fatigue, anxiety/sleep domains, while higher scores indicate better health for the physical function and satisfaction domains. The single Pain Intensity item is scored 0 (No pain) to 10 (Worst imaginable pain) in the past 7 days.
  Further details on PROMIS scoring are available at https://www.healthmeasures.net/images/PROMIS/manuals/PROMIS_Adult_Profile_Scoring_Manual.pdf.
Time Frame: 4, 8, and 12 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 135 | 135
score on a scale
  Physical Function: 4 month: number analyzed (Participants) | 121 | 122
  Physical Function: 4 month | 41.4 [35.8 to 47.6] | 41.8 [36.9 to 56.9]
  Physical Function: 8 month: number analyzed (Participants) | 117 | 121
  Physical Function: 8 month | 41.9 [37.6 to 56.9] | 42.1 [37.6 to 48.1]
  Physical Function: 12 month: number analyzed (Participants) | 119 | 119
  Physical Function: 12 month | 41.4 [36.4 to 48.2] | 41.7 [36.4 to 56.9]
  Depression and Sadness: 4 month: number analyzed (Participants) | 121 | 122
  Depression and Sadness: 4 month | 48.9 [41.0 to 55.5] | 41.0 [41.0 to 54.3]
  Depression and Sadness: 8 month: number analyzed (Participants) | 117 | 121
  Depression and Sadness: 8 month | 41.0 [41.0 to 53.0] | 41.0 [41.0 to 53.0]
  Depression and Sadness: 12 month: number analyzed (Participants) | 119 | 119
  Depression and Sadness: 12 month | 41.0 [41.0 to 55.5] | 41.0 [41.0 to 55.5]
  Pain Interference: 4 month: number analyzed (Participants) | 121 | 122
  Pain Interference: 4 month | 55.7 [41.6 to 61.3] | 54.85 [41.6 to 61.3]
  Pain Interference: 8 month: number analyzed (Participants) | 117 | 121
  Pain Interference: 8 month | 54.5 [41.6 to 60.0] | 54.4 [41.6 to 59.9]
  Pain Interference: 12 month: number analyzed (Participants) | 119 | 119
  Pain Interference: 12 month | 53.9 [41.6 to 61.3] | 53.9 [41.6 to 59.7]
  Ability to Participate: 4 month: number analyzed (Participants) | 121 | 122
  Ability to Participate: 4 month | 51.8 [45.0 to 58.3] | 48.3 [44.2 to 58.5]
  Ability to Participate: 8 month: number analyzed (Participants) | 117 | 121
  Ability to Participate: 8 month | 51.8 [44.2 to 58.1] | 51.8 [46.0 to 64.2]
  Ability to Participate: 12 month: number analyzed (Participants) | 119 | 119
  Ability to Participate: 12 month | 51.8 [44.6 to 58.3] | 51.7 [44.2 to 57.6]
  Fatigue: 4 month: number analyzed (Participants) | 121 | 122
  Fatigue: 4 month | 51.0 [46.4 to 59.3] | 53.1 [46.1 to 58.9]
  Fatigue: 8 month: number analyzed (Participants) | 117 | 121
  Fatigue: 8 month | 51.0 [46.4 to 57.1] | 51.0 [46.0 to 57.2]
  Fatigue: 12 month: number analyzed (Participants) | 119 | 119
  Fatigue: 12 month | 51.0 [46.0 to 57.1] | 51.3 [48.6 to 60.7]
  Anxiety and Fear: 4 month: number analyzed (Participants) | 121 | 122
  Anxiety and Fear: 4 month | 48.1 [40.3 to 57.5] | 48.8 [40.3 to 56.0]
  Anxiety and Fear: 8 month: number analyzed (Participants) | 117 | 121
  Anxiety and Fear: 8 month | 48.1 [40.3 to 55.6] | 47.9 [40.3 to 56.0]
  Anxiety and Fear: 12 month: number analyzed (Participants) | 119 | 119
  Anxiety and Fear: 12 month | 48.1 [40.3 to 56.0] | 47.9 [40.3 to 56.0]
  Sleep Disturbance: 4 month: number analyzed (Participants) | 121 | 122
  Sleep Disturbance: 4 month | 51.4 [43.8 to 55.8] | 51.1 [44.2 to 54.5]
  Sleep Disturbance: 8 month: number analyzed (Participants) | 117 | 121
  Sleep Disturbance: 8 month | 51.1 [45.3 to 54.7] | 51.0 [43.5 to 55.3]
  Sleep Disturbance: 12 month: number analyzed (Participants) | 119 | 119
  Sleep Disturbance: 12 month | 51.1 [44.6 to 55.5] | 51.7 [45.1 to 55.5]
  Pain Intensity: 4 month: number analyzed (Participants) | 121 | 122
  Pain Intensity: 4 month | 3 [1 to 5] | 2 [1 to 5]
  Pain Intensity: 8 month: number analyzed (Participants) | 117 | 121
  Pain Intensity: 8 month | 2 [1 to 4] | 2 [0 to 5]
  Pain Intensity: 12 month: number analyzed (Participants) | 119 | 119
  Pain Intensity: 12 month | 3 [0 to 5] | 3 [0 to 5]

5. Secondary Outcome: Emergency Room Visits
Description: The number of participants with 1 or more emergency room visits will be quantified at 12 months. Data will be used to compare health care utilization between the two study arms.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: Receive a brochure on atrial fibrillation that is published by the American Heart Association and a smartphone with the WebMD application.
  Participants are directed to use the WebMD application as often as they would like.
  Usual Care: Use of the WebMD app daily for 120 days.
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 135 | 135
Participants
  Participants with no ER visits | 92 | 92
  Participants with 1 or more ER visits | 43 | 43

6. Secondary Outcome: Hospital Admissions
Description: The number of participants with one or more hospitalization will be quantified at 12 months. Data will be used to compare health care utilization between the two study arms.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 135 | 135
Participants
  Participants with no hospital admission | 99 | 103
  Participants with 1 or more hospital admissions | 36 | 32

ADVERSE EVENTS:
Time Frame: Data collection occurred from date of consent through the participants 12-month visit.
Description: The study team will learn of adverse events (AE) and serious AEs (SAE) by participant interview at the 4-, 8-, and 12-month assessments; direct contact by participants during the scheduled check-in calls; review of the electronic health record; communication from referring physicians or participants'' providers; or contact with study team initiated by family or other participant surrogates.
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/135 | 6/135
Serious Adverse Events (participants affected / at risk) | 35/135 | 31/135
Other Adverse Events (participants affected / at risk) | 32/135 | 40/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=135) | Usual Care (N=135)
Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 12 (12) | 0 (0)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0)
Heart failure (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Other (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary duct inflamation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestine obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other (Gastrointestinal disorders) | 2 (2) | 0 (0)
Death NOS (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
COVID-19 (General disorders) | 1 (1) | 0 (0)
Other (General disorders) | 1 (1) | 0 (0)
Cholecystitis (General disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (2)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 5 (7)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (2) | 3 (4)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=135) | Usual Care (N=135)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (6) | 4 (4)
Chest pain-cardiac (Cardiac disorders) | 2 (3) | 3 (4)
Heart Failure (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other (Gastrointestinal disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2)
COVID-19 (General disorders) | 1 (1) | 2 (2)
Other (General disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (7) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other (Injury, poisoning and procedural complications) | 2 (2) | 6 (7)
INR increased (Investigations) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Other (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other (Surgical and medical procedures) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 1 (1)
Unknown classification (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT04076020/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT04076020/ICF_001.pdf